CLINICAL TRIAL: NCT05204823
Title: Evaluation of the Glycemic Index in 4 Dairy Beverages.
Acronym: IG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-00023
Record Dates: First submitted 2021-12-22; First posted 2022-01-24 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2021-11

CONDITIONS: Glycemic Index; Cognitive Performance
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental Product 1 (Experimental): Consumption of 221.24 ml of product 1 (corresponding to 25g of glucose). Subjects will take this amount only on the day of the visit that they are to consume this product.
  Interventions: Other: Experimental product
- Experimental Product 2 (Experimental): Consumption of 282.81 ml of product 1 (corresponding to 25g of glucose). Subjects will take this amount only on the day of the visit that they are to consume this product.
  Interventions: Other: Experimental product
- Experimental Product 3 (Experimental): Consumption of 589,62 ml of product 1 (corresponding to 25g of glucose). Subjects will take this amount only on the day of the visit that they are to consume this product.
  Interventions: Other: Experimental product
- Experimental Product 4 (Experimental): Consumption of 573,39 ml of product 1 (corresponding to 25g of glucose). Subjects will take this amount only on the day of the visit that they are to consume this product.
  Interventions: Other: Experimental product
- Control product (Active Comparator): Consumption of 25g of glucose. Subjects will take this amount only on the day of the visit that they are to consume this product.
  Interventions: Other: Control product

INTERVENTIONS:
Other: Experimental product — Chocolate milk shakes
  Arms: Experimental Product 1; Experimental Product 2; Experimental Product 3; Experimental Product 4
Other: Control product — Glucose
  Arms: Control product

SUMMARY:
The objective of the study is to evaluate the glycemic index and glycemic load of 4 chocolate milk drinks.

DETAILED DESCRIPTION:
Subjects will make a total of 5 visits. Four visits where they will drink a chocolate milkshake at each visit. In the other visit they will take glucose, as a comparator product.

Due to the low amount of sugars in the shakes, subjects will drink the equivalent of 25g of glucose.

At each visit subjects will have to come fasting, and samples will be collected at 9 different times.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes (10 men and 10 women).
* Subjects aged between 20 and 35 years.
* Subjects with a body mass index between 20 and 25 kg/m2.

Exclusion Criteria:

* Subjects suffering from diabetes mellitus or any chronic disease.
* Subjects with medical problems or a diagnosed psychiatric disorder.
* Subjects with alcohol abuse or excessive alcohol consumption (>3 glasses of wine or beer/day).
* Subjects consuming any pharmacological medication that may affect memory.
* Participation in another clinical trial in the three months prior to the study.
* Unwillingness or inability to comply with clinical trial procedures.
* Subjects whose condition does not make them eligible for the study according to the investigator's criteria.
* Pregnant or lactating women.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Glucose | The glucose evolution will be measured for 210 minutes after product consumption.
  It will be evaluated by means of a glucometer.

SECONDARY OUTCOMES:
Glucose | Each product will be measured at 15, 30, 45, 60, 90, 120 and 150 minutes after consumption.
  It will be evaluated by means of a glucometer.

CONTACTS AND LOCATIONS:
Overall Officials: Fco Javier López Román, Principal Investigator — Catholic University of Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain